CLINICAL TRIAL: NCT06753422
Title: Effects of Kefir Consumption on Gut Microbiota and Athletic Performance in Professional Female Soccer Players: a Randomized Controlled Trial
Brief Title: Kefir, Gut Microbiota, and Athletic Performance in Soccer Players
Acronym: KEFIR-SPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-KefirStudy; TDK-2023-91 (Other Grant/Funding Number: Acıbadem University Scientific Research Projects Unit (BAP))
Record Dates: First submitted 2024-12-20; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Gut Microbiota Diversity and Composition; Athletic Performance; Functional Food Intervention (Kefir); Body Composition; Dietary Intake Patterns
Keywords: Kefir; Gut microbiota; Athletic performance; Female Athletes; Functional foods; Body composition; Dietary intake
MeSH Terms: interventions — Kefir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kefir Consumption Group (Experimental): Participants in this group will consume 200 ml of kefir daily for 4 weeks. Their diet will remain ad libitum, with no additional dietary restrictions or standardization applied during the intervention period.
  The primary intervention in our study is the daily consumption of kefir (200 ml/day). No additional drug or medical device was used during the intervention or data collection process. The study focused solely on kefir consumption and its effects on athletic performance and gut microbiota.
  Interventions: Dietary Supplement: Kefir
- Control Group (No Intervention): Participants in this group will not receive any specific intervention. They will continue their usual diet ad libitum, with no dietary restrictions or standardization applied during the study period.

INTERVENTIONS:
Dietary Supplement: Kefir — 200 ml/day kefir
  The primary intervention in our study is the daily consumption of kefir (200 ml/day). No additional drug or medical device was used during the intervention or data collection process. The study focused solely on kefir consumption and its effects on athletic performance and gut microbiota.
  Other Names: Altınkılıç Lactose-free Kefir, The kefir product used in this study was purchased independently with no sponsorship or involvement from the manufacturer
  Arms: Kefir Consumption Group

SUMMARY:
This research work is a clinical trial that will assess the impact of kefir consumption on the gut microbiota profile and athletic performance of female soccer players of age 18-29 years. The participants were divided into two groups namely the kefir intervention group and the control group. The primary end points are the modifications in the alpha diversity of the gut microbiome and the beta diversity of the gut microbiome and also the athletic performance outcomes like VO2 max and finishing speed which will be measured using the 30-15 Intermittent Fitness Test. The other outcomes of the study are the changes in the body composition (measured through BIA and skinfold), the changes in the dietary intake and the variations in certain microbial genera such as Akkermansia muciniphila and Faecalibacterium prausnitzii.

The study will be the first to evaluate whether kefir intake can increase the microbial diversity, increase the VO2max and improve the body composition of professional athletes. The anticipated outcomes of this study are enhanced gut microbial diversity, enhanced VO2max and finishing speed, and positive alteration in the body composition parameters.

DETAILED DESCRIPTION:
This randomized controlled trial aims at evaluating the impact of kefir on the participants' gut microbiota and athletic performance among professional female soccer players of 18-29 years. The present study is intended to reveal the potential of kefir, a fermented milk product that is packed with probiotics , in altering the diversity and profile of gut microbiota, physical performance, and parameters of body composition.

This trial was carried out for a period of four weeks and the subjects were divided into two parallel groups; the kefir group in which the participants consume 200ml of kefir per day and the control group in which the participants continued with their normal diet without kefir supplementation. The subjects were assigned to either of the two groups at the beginning of the study. Since the study involved a dietary intervention, the trial was conducted without blinding the subject and the researcher. Measurements were made at the beginning and at the end of the intervention in order to evaluate the outcomes.

The main goals of the study were to observe the changes in the diversity and the composition of the gut microbiome with the help of 16S rRNA sequencing and to determine the changes in the athletic performance indices including VO2max and finishing speed which was measured by 30-15 Intermittent Fitness Test. Other objectives were to establish the effects of kefir on other body composition measures such as body fat percentage, fat free mass and total body weight , to examine the patterns of dietary intakes and their relationships with the microbiota and performance measures and to examine the changes in certain gut microorganisms including Akkermansia muciniphila and Faecalibacterium prausnitzii which are known to have positive effects on human health and performance.

The alpha diversity of the gut microbiome was measured with the Shannon and Chao1 indices and the beta diversity was calculated with the Bray-Curtis dissimilarity. The taxonomic analysis was done at the phylum, genus and species level in order to identify the changes in the microbial community due to consumption of kefir. The participants' athletic performance was evaluated with IFT Test to explore the changes in VO2max and finishing speed. Changes in the body composition were assessed by Bioelectrical Impedance Analysis (BIA) and skinfold callipers and the dietary intake data were collected through three-day food records, one off day and two training days to examine the macronutrients and micronutrients intake and their relationship with the microbiota and performance.

This trial seeks to fill an important research gap in the current literature on functional foods in sports nutrition with focus on professional female athletes. In this way, the current study seeks to link dietary interventions with the gut microbiota as well as performance parameters in order to provide empirical support for how kefir can improve the gut health and performance of athletes and to facilitate the development of personalised nutrition for athletes.

ELIGIBILITY:
Inclusion criteria:

* Professional female soccer player
* Aged between 18 and 35 years
* Regular participation in a structured training program
* No allergy or intolerance to kefir or dairy products
* Willingness to voluntarily participate in the study
* Signed informed consent form

Exclusion criteria:

* History of allergy or intolerance to kefir or dairy products
* Presence of chronic diseases (e.g., diabetes, heart disease, kidney failure)
* Use of antibiotics or probiotic supplements within the last 3 months
* Pregnancy or breastfeeding
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota Composition Change | At baseline and after 4 weeks of intervention (Week 5)
  Changes in gut microbiota diversity and abundance at genus and phylum levels, assessed through 16S rRNA gene sequencing of stool samples.
Athletic Performance Improvement | At baseline and after 4 weeks of intervention (Week 5)
  Improvement in athletic performance as measured by the 30-15 Intermittent Fitness Test, evaluating VO2max and finishing speed.

SECONDARY OUTCOMES:
Dietary Intake Assessment | At baseline and after 4 weeks of intervention (Week 5)
  Changes in macronutrient and micronutrient intake, assessed through 3-day food records analyzed using nutritional analysis software (BEBIS).
Body weight (kg) | At baseline and after 4 weeks of intervention (Week 5)
  Body weight will be measured using a bioelectrical impedance analysis (BIA) device (Tanita BC 545-N ) to assess participants' total body weight.
Body Fat Percentage (%) | At baseline and after 4 weeks of intervention (Week 5)
  Body fat percentage will be measured using a bioelectrical impedance analysis (BIA) device (Tanita BC 545-N ) to assess the proportion of body weight composed of fat tissue.
Fat mass (kg) | At baseline and after 4 weeks of intervention (Week 5)
  Fat mass will be measured using a bioelectrical impedance analysis (BIA) device (Tanita BC 545-N ) to quantify the total weight of fat tissue in the body.
Fat-free mass (kg) | At baseline and after 4 weeks of intervention (Week 5)
  Fat-free mass will be measured using a bioelectrical impedance analysis (BIA) device (Tanita BC 545-N ) to determine the weight of lean tissue, bones, and fluids, excluding fat mass.
Height (m) | At baseline and after 4 weeks of intervention (Week 5)
  Height will be measured using a SECA 213 stadiometer with participants standing upright, without shoes, and with their head in the Frankfurt plane.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sağlam, Associate Professor, Study Chair — Acibadem University
Locations (1):
- Fatih Vatan Sports Club, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from gut microbiota analysis, including genus and phylum-level diversity and abundance, assessed using 16S rRNA sequencing.
  De-identified performance test data, such as VO2max and finishing speed results from the 30-15 Intermittent Fitness Test.
  De-identified body composition data, including body fat percentage and lean muscle mass assessed using BIA and caliper measurements.
  De-identified dietary intake data collected through 3-day food records, including macronutrient and micronutrient consumption.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD and supporting documents (e.g., Study Protocol, SAP) will be available starting 6 months after publication of primary results and will remain available indefinitely
Access Criteria: Researchers with a methodologically sound research proposal, approved by an independent ethics committee, will be able to access de-identified individual participant data (IPD) and supporting documents (e.g., Study Protocol, SAP). Data will be shared through a secure online repository upon request. Access will be granted after signing a Data Use Agreement, ensuring data confidentiality and ethical use.